CLINICAL TRIAL: NCT01927783
Title: Cardiovascular Health and Needs Assessment in Washington D.C. - Development of a Community-Based Behavioral Weight Loss Intervention
Brief Title: Heart Health Study in Washington D.C. to Develop a Community-Based Behavioral Weight Loss Intervention
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130183; 13-H-0183
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12-29

CONDITIONS: Cardiovascular Disease; Obesity
Keywords: Cardiovascular Disease; Obesity; Natural History
MeSH Terms: conditions — Cardiovascular Diseases; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1: Healthy Volunteer
- Group 2: Focus Group- Neighborhood and Physical Activity
- Group 3: Focus Group
- Group 4: Focus Group- Mobile App
- Group 5: Consent for Cooking Survey Focus Group
- Group 6: Community Organization Survey focus Group

SUMMARY:
Background:

- Past studies suggest that the best way to improve heart health in the Black community is through community-based programs. Researchers will partner with DC community leaders. They will collect information about the health and health needs of people in mostly Black churches in DC. They will study things that affect heart health, like diabetes, blood pressure, cholesterol, and weight. They will also study how technology can keep track of activities and health. The information will show the health needs of church-based communities or faith-based organizations.

Objectives:

- The primary objective of this study is to estimate the percentage of the population that meet ideal, intermediate, and poor criteria for each of the cardiovascular health factors (BMI, physical activity, dietary intake, blood pressure, total cholesterol, fasting plasma glucose, and cigarette smoking) in churches or faith-based organizations in the DMV area. This data will inform the design and implementation of a behavioral weight-loss intervention within the faith-based community immediately following this study.

The secondary objectives are to: 1) evaluate usage of handheld devices for objectively measuring physical activity and dietary intake; 2) evaluate usage of web-based technology for monitoring cardiovascular health markers, including dietary intake; 3) examine referral methods for untreated hypertension, diabetes, and hypercholesterolemia; 4) compare lifestyle behaviors across levels of psychosocial factors, cultural norms, and neighborhood environment factors; and 5) formalize a community advisory board involved in the implementation of the health screening and needs assessment program and a future behavioral weight-loss intervention.

Eligibility:

- Adults ages 19 to 85 who attend one of the study churches.

Design:

* Participants will visit their church for a 4-hour health exam. They will have their blood pressure and body measurements taken. They will have a drop of blood taken from their finger with a small needle. This blood will be tested for blood sugar and cholesterol. Participants will be given the results of these tests.
* Participants will answer questions about their health.
* All participants will be given an activity monitor to wear for 1 month. The activity monitor is worn around the wrist. Some participants will also receive an activity monitor that is worn around the waist. Participants will be given instructions on how to wear the activity monitors and follow the results on a website.
* At the end of 1 month, participants will return one device (they can keep the other). They may receive a gift card for completing the study.

DETAILED DESCRIPTION:
Obesity leads to an increased risk of cardiovascular risk factors and death from cardiovascular disease. Therefore, interventions that slow or reverse the obesity epidemic are essential. Community-based interventions can reach those most at risk for obesity and obesity-related cardiovascular risk factors. Interventions based on community-based participatory research (CBPR) principles develop in collaboration with community partners, allowing an intervention s components to be tailored to the unique needs of the community members. To remain consistent with CBPR principles, a community assessment is necessary to understand the needs of the target population. Therefore, we propose a cardiovascular health screening and needs assessment of a sample population from churches or faith-based organizations in DC, Maryland, and Virginia where obesity prevalence is highest and resources for physical activity and healthy nutrition are most limited. The screening will involve measuring cardiovascular health factors such as body mass index (BMI), physical activity, dietary intake, total cholesterol, blood pressure, fasting plasma glucose, and cigarette smoking. Based on American Heart Association-established goals, cardiovascular health factors can be defined as ideal, intermediate, or poor, depending on control of risk factors and lifestyle behaviors. In this protocol, we will determine the prevalence of ideal, intermediate, and poor cardiovascular health factors within the church or faith-based organization population. We hypothesize that the percentage of the church or faith-based organization population that meets ideal criteria for each of the cardiovascular health factors will be lower than the percentage meeting intermediate and poor criteria for the cardiovascular health factors. In addition, we will evaluate the use of handheld technology for objectively measuring physical activity and the use of web-based technology for monitoring cardiovascular health factors within the population. We will also evaluate social determinants of health, particularly psychosocial and environmental factors that might hinder weight loss. Finally, we will establish a community advisory board to consult on the planning and implementation of the assessment, and the interpretation and dissemination of study findings. The results of this community-based, cardiovascular health and needs assessment will inform the design and implementation of a future community-based behavioral weight loss intervention.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals eligible for this protocol are aged 19 - 85 years, have attended or visited any church or faith-based organization in DC, Maryland, or Virginia, and are able to provide informed consent independently. Eligible participants should also speak and read English at the 8th grade level.

EXCLUSION CRITERIA:

Women in their second or third trimester of pregnancy at the time of enrollment will be excluded from the protocol.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This observational study will may involve cardiovascular health factor screening, administration of a survey, and evaluating usage of handheld and web-based technology related to physical activity, dietary intake, and cardiovascular health for one-month intervals through the duration of the study (for a maximum of 6 months) for a convenience sample of participants recruited from churches in Wards 5, 7, or 8 in Washington D.C and in neighboring Prince George s County.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-02-08 (Actual); Primary Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
estimate CVD risk factors in Ward 5,7,8 | ongoing
  data will inform the design and implementation of a behavioral weight-loss intervention within the faith-based community immediately following this study

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany M Powell-Wiley, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available

REFERENCES:
- [Derived] Claudel SE, Tamura K, Troendle J, Andrews MR, Ceasar JN, Mitchell VM, Vijayakumar N, Powell-Wiley TM. Comparing Methods to Identify Wear-Time Intervals for Physical Activity With the Fitbit Charge 2. J Aging Phys Act. 2021 Jun 1;29(3):529-535. doi: 10.1123/japa.2020-0059. Epub 2020 Dec 16. PMID 33326935
- [Derived] Fowler LA, Yingling LR, Brooks AT, Wallen GR, Peters-Lawrence M, McClurkin M, Wiley KL Jr, Mitchell VM, Johnson TD, Curry KE, Johnson AA, Graham AP, Graham LA, Powell-Wiley TM. Digital Food Records in Community-Based Interventions: Mixed-Methods Pilot Study. JMIR Mhealth Uhealth. 2018 Jul 17;6(7):e160. doi: 10.2196/mhealth.9729. PMID 30021705
- [Derived] Yingling LR, Brooks AT, Wallen GR, Peters-Lawrence M, McClurkin M, Cooper-McCann R, Wiley KL Jr, Mitchell V, Saygbe JN, Johnson TD, Curry RK, Johnson AA, Graham AP, Graham LA, Powell-Wiley TM. Community Engagement to Optimize the Use of Web-Based and Wearable Technology in a Cardiovascular Health and Needs Assessment Study: A Mixed Methods Approach. JMIR Mhealth Uhealth. 2016 Apr 25;4(2):e38. doi: 10.2196/mhealth.4489. PMID 27113680
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-H-0183.html